CLINICAL TRIAL: NCT05450770
Title: The Yellow Fever Vaccine Immunity in HIV Infected Patients: Studies of Immunological Responses at 10 Years (ANRS 0146s NovaaTen)
Brief Title: Immunity to Yellow Fever in HIV-infected Patients 10 Years After a Primary Anti-yellow Fever Vaccination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Saint-Louis Hospital, Paris, France (Other); Bichat Hospital (Other); Hôpital Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 0146s NovaaTen
Record Dates: First submitted 2022-06-14; First posted 2022-07-11 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; Yellow Fever
MeSH Terms: conditions — HIV Infections; Yellow Fever

STUDY DESIGN:
Intervention Model Description: Category 2, multi-centric intervention research comparing 2 parallel groups of 40 HIV + subjects and 20 HIV- subjects included in the ANRS EP46 NOVAA trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV+ GROUP (Active Comparator): Subjects included in the ANRS EP 46 NOVAA trial:
  • 40 HIV positive subjects from consultations for infectious diseases and travel medicine centers at Saint-Louis, Cochin-Pasteur and Bichat hospitals (on HAART for at least one year and not modified in the 3 months preceding the pre-inclusion visit, CD4 > 350/mm3 and a viral load <50 copies / mL for at least 6 months).
  Interventions: Biological: Yellow fever vaccination (STAMARIL)
- HIV- GROUP (Other): Subjects included in the ANRS EP 46 NOVAA trial:
  • 20 HIV negative subjects from the consultation of travelers from Saint-Louis, Bichat and Cochin-Pasteur hospitals.
  Interventions: Biological: Yellow fever vaccination (STAMARIL)

INTERVENTIONS:
Biological: Yellow fever vaccination (STAMARIL) — Yellow fever vaccination (STAMARIL) for HIV positive and negative subjects

SUMMARY:
ANRS 0146s NovaaTen study aims to determine the vaccine responses in the participants of the ANRS EP46 Novaa trial 10 years after a primary anti-yellow fever vaccination

DETAILED DESCRIPTION:
The vaccine responses will be determined with the measurement of the neutralizing antibody titers using the neutralization tests PRNT and Pseudo type ACN 400 to M120 (ten years) in the participants of the ANRS EP 46 NOVAA trial, VIH+ and controls naïve to previous vaccination ten years after a primary anti-yellow fever vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in the ANRS EP 46 NOVAA trial:

  * 40 HIV positive subjects from consultations for infectious diseases and travel medicine centers at Saint-Louis, Cochin-Pasteur and Bichat hospitals (on HAART for at least one year and not modified in the 3 months preceding the pre-inclusion visit, CD4 > 350/mm3 and a viral load <50 copies / mL for at least 6 months).
  * 20 HIV negative subjects from the consultation of travelers from Saint-Louis, Bichat and Cochin-Pasteur hospitals.
  * Subjects agreeing to be monitored according to the terms of the protocol.
  * Subjects affiliated to a Social Security scheme or beneficiaries of such a scheme.
  * Signature of informed consent.

Exclusion Criteria:

* Non-volunteers for the 10-year follow-up
* Subject under curatorship, guardianship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Immuno-virologic criterion | At Months 120 (10years)
  At Months 120 (10years), the antibody titers of neutralizers by PRNT (Plaque reduction neutralization test) and pseudotypes will be determined

SECONDARY OUTCOMES:
Predicting a sustained vaccine response 10 years later. | At Months 120 (10years)
  To study the effect of clinical and biological factors in HIV+ patients (collection of data on: age; clinical examination; heart rate; weight; body temperature; blood pressure; CD4, CD8 and the CD4/CD8 ratio; the nadir and zenith of CD4; the duration of antiretroviral treatment; the duration of HIV infection) on the PRNT titers transformed into logarithm and the percentages of neutralization at ten years, uni and multivariate regressions are used.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie COLIN de VERDIERE, Study Director — Maladies Infectieuses St Louis Paris; Odile LAUNAY, Principal Investigator — CIC Cochin Paris; Jade GHOSN, Principal Investigator — Hôpital Bichat Paris